CLINICAL TRIAL: NCT03560323
Title: Ketones, Muscle Metabolism, and SGLT2 Inhibitors - Protocol 1.
Acronym: Protocol1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20180077H; 2R01DK107680-06A1 (NIH)
Record Dates: First submitted 2018-06-04; First posted 2018-06-18 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Type 2 Diabetes Mellitus
Keywords: Ketone Body Metabolism; Myocardial Glucose Uptake; Positron Emission Tomography; Myocardial Function
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Type 2 diabetic subjects with New York Heart Association (NYHA) Class II-III heart failure and ejection fraction <50% (documented by patient's medical records with an Echocardiogram (ECHO) or any other heart imaging) will be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I Beta-Hydroxy-Butyrate (Active Comparator): Administration of beta-hydroxy-butyrate at 0.4 mg/kg.min for 20 minutes and then at a constant rate of 0.2 mg/kg.min until study end
  Interventions: Drug: Beta-hydroxy-butyrate
- Group II Beta-Hydroxy-Butyrate (Active Comparator): Administration of beta-hydroxy-butyrate at 1.5 mg/kg.min for 20 minutes and then at a constant rate of 0.75 mg/kg.min until study end
  Interventions: Drug: Beta-hydroxy-butyrate
- Group III Beta-Hydroxy-Butyrate (Active Comparator): Administration of beta-hydroxy-butyrate at 4.0 mg/kg.min for 20 minutes and then at a constant rate of 2.0 mg/kg.min until study end
  Interventions: Drug: Beta-hydroxy-butyrate

INTERVENTIONS:
Drug: Beta-hydroxy-butyrate — Following completion of the baseline MRI and blood samples, subjects will be divided into three groups (26 subjects per group). Each group will receive a 6-hour (3-hour in group III) prime-continuous infusion of racemic B-OH-B (100 mg/mL solution; pH adjusted to 7.4) to increase the plasma B-OH-B concentration by 0.5, 2.0, and 5.0 mmol/L.
  GROUP I: Prime = 0.4 mg/kg.min for 20 minutes and constant rate = 0.2 mg/kg.min until study end GROUP II: Prime = 1.5 mg/kg.min for 20 minutes and constant rate = 0.75 mg/kg.min until study end GROUP III: Prime = 4.0 mg/kg.min for 20 minutes and constant rate = 2.0 mg/kg.min until study end
  Other Names: Infusion of Beta-Hydroxy-Butyrate (B-OH-B)

SUMMARY:
To examine the effect of an increase in plasma beta-hydroxy-butyrate (B-OH-B) levels, spanning the physiologic and pharmacologic range (+0.5, +2.0, and +5.0 mmol/L), on: (i) parameters of left ventricular (LV) systolic and diastolic function utilizing cardiac magnetic resonance imaging (MRI) and (ii) myocardial glucose uptake using positron emission tomography (PET) with 18F-fluoro-2-deoxy-D-glucose in type 2 diabetic patients with Class II-III New York Heart Association (NYHA).

DETAILED DESCRIPTION:
Purpose/Objectives The EMPA-REG OUTCOME (NCT01131676) trial demonstrated that SGLT2 (sodium-glucose co-transporter) inhibition with empagliflozin markedly reduced cardiovascular (CV) mortality and hospitalization for heart failure. In diabetic patients treated with SGLT2 inhibitors, a rise in plasma ketone concentration consistently has been observed. This has led to the "ketone hypothesis" in which a shift from glucose/FFA (Free Fatty Acids) to ketone utilization by the heart results in enhanced left ventricular systolic/diastolic function and could, at least in part, explain the reduction in CV mortality and hospitalization for heart failure observed in the EMPA-REG OUTCOME trial.

Methods Type 2 diabetic subjects with New York Heart Association (NYHA) Class II-III heart failure and ejection fraction less than 50% will be studied. Eligible subjects will undergo a baseline cardiac MRI to obtain quantitative measures of baseline cardiac functional parameters: chamber volumes and pressures, wall thickness, LV diastolic function (E/A ratio, peak LV filling rate, diastolic volume), LV systolic function (cardiac output, stroke volume, systolic volume, peak LV ejection rate). Baseline samples will be drawn for measurement of N-terminal pro-brain natriuretic peptide (NT-proBNP) , B-OH-butyrate, acetoacetate, glucose, FFA, lactate, pyruvate, glycerol, HCO3 (bicarbonate), insulin, glucagon, renin and aldosterone. Following completion of the baseline MRI and blood samples, subjects will be divided into three groups (12 subjects per group). Each group will receive a 6-hour (3-hour in group III) prime-continuous infusion of racemic B-OH-B (100 mg/mL solution; pH adjusted to 7.4) to increase the plasma B-OH-B concentration by ~0.5, ~2.0, and ~5.0 mmol/L. At the end of the infusion the MRI will be repeated. As a time control GROUP II subjects will receive a continuous infusion of sodium bicarbonate (0.12 M) for 6 hours (0.08 mg/kg/min) to mimic the rise in plasma bicarbonate concentration observed with B-OH-B infusion. Group II will return again to the RII (UT Health Research Imaging Institute) on a separate day for a cardiac positron emission tomography (PET) study to examine the effect of hyperketonemia on myocardial glucose uptake and blood flow. In ~14 days subjects will return for a repeat PET/18F-2-DOG (deoxyglucose) study with one exception: NaHCO3 (Sodium bicarbonate) will be infused instead of B-OH-B. The two studies will be performed in random order.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes.
2. Class II-III New York Heart Association (NYHA) heart failure with ejection fraction less than 50 %.
3. Age 18-80 years.
4. BMI 23-38 kg/m2.
5. HbA1c 6.0-9.0 %.
6. Blood pressure < 145/85 mmHg.
7. eGFR > 30 mL/min/1.73 m2.
8. NT-proBNP ≥ 500 pg/mL (or ≥ 300 pg/mL if ejection fraction is less than 35 %).

Exclusion Criteria:

1. Treatment with Glucagon-like peptide-1 receptor agonist (GLP-1 RA), Dipeptidyl peptidase-4 inhibitors (DPP4i), pioglitazone, SGLT2 inhibitor or insulin.
2. Women who are pregnant or breastfeeding.
3. Contraindications for MRI include metal plates, parts, screws, shrapnel, pins in the body, or cardiac pacemaker.
4. Any other condition that in the opinion of the investigator create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — UT Health San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I Beta-Hydroxy-Butyrate: Administration of beta-hydroxy-butyrate at 0.4 mg/kg.min for 20 minutes and then at a constant rate of 0.2 mg/kg.min until study end
  Beta-hydroxy-butyrate: Following completion of the baseline MRI and blood samples, subjects will be divided into three groups (26 subjects per group). Each group will receive a 6-hour (3-hour in group III) prime-continuous infusion of racemic B-OH-B (100 mg/mL solution; pH adjusted to 7.4) to increase the plasma B-OH-B concentration by 0.5, 2.0, and 5.0 mmol/L.
  GROUP I: Prime = 0.4 mg/kg.min for 20 minutes and constant rate = 0.2 mg/kg.min until study end GROUP II: Prime = 1.5 mg/kg.min for 20 minutes and constant rate = 0.75 mg/kg.min until study end GROUP III: Prime = 4.0 mg/kg.min for 20 minutes and constant rate = 2.0 mg/kg.min until study end
- Group II Beta-Hydroxy-Butyrate: Administration of beta-hydroxy-butyrate at 1.5 mg/kg.min for 20 minutes and then at a constant rate of 0.75 mg/kg.min until study end
  Beta-hydroxy-butyrate: Following completion of the baseline MRI and blood samples, subjects will be divided into three groups (26 subjects per group). Each group will receive a 6-hour (3-hour in group III) prime-continuous infusion of racemic B-OH-B (100 mg/mL solution; pH adjusted to 7.4) to increase the plasma B-OH-B concentration by 0.5, 2.0, and 5.0 mmol/L.
  GROUP I: Prime = 0.4 mg/kg.min for 20 minutes and constant rate = 0.2 mg/kg.min until study end GROUP II: Prime = 1.5 mg/kg.min for 20 minutes and constant rate = 0.75 mg/kg.min until study end GROUP III: Prime = 4.0 mg/kg.min for 20 minutes and constant rate = 2.0 mg/kg.min until study end
- Group III Beta-Hydroxy-Butyrate: Administration of beta-hydroxy-butyrate at 4.0 mg/kg.min for 20 minutes and then at a constant rate of 2.0 mg/kg.min until study end
  Beta-hydroxy-butyrate: Following completion of the baseline MRI and blood samples, subjects will be divided into three groups (26 subjects per group). Each group will receive a 6-hour (3-hour in group III) prime-continuous infusion of racemic B-OH-B (100 mg/mL solution; pH adjusted to 7.4) to increase the plasma B-OH-B concentration by 0.5, 2.0, and 5.0 mmol/L.
  GROUP I: Prime = 0.4 mg/kg.min for 20 minutes and constant rate = 0.2 mg/kg.min until study end GROUP II: Prime = 1.5 mg/kg.min for 20 minutes and constant rate = 0.75 mg/kg.min until study end GROUP III: Prime = 4.0 mg/kg.min for 20 minutes and constant rate = 2.0 mg/kg.min until study end
Period: Overall Study
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Started | 13 | 14 | 13
Completed | 12 | 12 | 12
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants were recruited from the Heart Failure (HF) clinic of UT Health San Antonio and from the Texas Diabetes Institute. Before the screening visit, patients had an established diagnosis of HF documented by an acceptable imaging modality within 6 months.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate | Total
Number analyzed (Participants) | 13 | 14 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 12 | 35
  >=65 years | 1 | 3 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (2) | 60 (2) | 57 (3) | 58 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 12 | 11 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 8 | 28
  Not Hispanic or Latino | 3 | 4 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 13 | 13 | 10 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output (CO)
Description: Within 2 weeks after the screening visit, subjects return to the Research Institute (RII) at 7:00AM for a cardiac MRI on 3.0T MRI System (TIM, Trio, Siemens Medical Solution, Malvern, PA).
  Cardiac output (CO) is measured using velocity encoded phase contrast MRI. The patient lies in the MRI scanner, and the imaging plane is positioned perpendicular to the ascending aorta where blood flow can be measured accurately. The MRI scan is synchronized with the patient's heartbeats using ECG gating. Two types of images are collected: magnitude images, which provide anatomical reference, phase images, which encode the speed and direction of blood flow. The system multiplies velocity by the cross-sectional area of the vessel to calculate the volume of blood passing through the vessel at each moment. Integrating the flow values over the entire cardiac cycle, the system calculates the stroke volume. Cardiac Output = Stroke Volume × Heart Rate
Time Frame: Baseline at 0 minute before B-OH-B infusion and 360 minutes after B-OH-B infusion for Group I & II. For Group III was baseline at 0 minute and 180 minutes after infusion
Population: Patients with diabetes who met entry criteria were randomized (1:1:1 ratio) to receive one of three different infusion rates of b-OH-B ((prime dose was 0.4 mg/kg/min for 20 min followed by constant rate of infusion 0.2 mg/kg/min until study end). Group I and Group II received a 6-h b-OH-B infusion. Group III received a 3-h b-OH-B infusion
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Number analyzed (Participants) | 12 | 12 | 12
mL/min
  Baseline:before Beta-H-B infusion infusion | 5.02 (0.38) | 4.54 (0.28) | 5.93 (0.36)
  After Beta-H-B infusion infusion | 5.10 (0.41) | 5.3 (0.22) | 7.16 (0.44)

2. Primary Outcome: Ejection Fraction (EF)
Description: A measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each heartbeat. It's a key indicator of heart function and can help diagnose and track heart failure. A normal EF typically falls between 55% and 70%. Values below 40% are often considered indicative of heart failure.
Time Frame: Baseline at 0 minute before infusion and 360 minutes after infusion for Group I & II. Group III was baseline at 0 minute of infusion and 180 minutes after infusion
Population: Below showed the difference before and after infusion. Patients were randomized (1:1:1 ratio) to receive one of three different infusion rates of b-OH-B ((prime dose was 0.4 mg/kg/min for 20 min followed by constant rate of infusion 0.2 mg/kg/min until study end). Group I and Group II received a 6-h b-OH-B infusion. Group III received a 3-h b-OH-B infusion
Measure: Mean (Standard Deviation); unit: percentage(%)
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Number analyzed (Participants) | 12 | 12 | 12
percentage(%) | 0.1 (1.2) | 3.9 (3.5) | 6.4 (4.5)

3. Primary Outcome: Left Ventricular Stroke Volume (LVSV)
Description: Represents the amount of blood ejected from the heart's left ventricle with each heartbeat. It's a crucial indicator of cardiac function, reflecting how effectively the heart pumps blood to the body.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mL/m²
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Number analyzed (Participants) | 12 | 12 | 12
mL/m² | 0.3 (1.3) | 9.7 (6.4) | 19.4 (6.0)

4. Secondary Outcome: Myocardial Energetics-Myocardial Glucose Uptake (MGU)
Description: A sub-set of participants in group II also underwent a cardiac PET study to examine the effect of hyperketonemia on Myocardial Glucose Uptake (MGU) and Myocardial Blood Flow MBF). A 20-min transmission scan was performed after exposure to a retractable 68Ge ring source to correct emission data for tissue attenuation of g photons. Then, 15O-H2O (10.5 MBq/kg) was administered intravenously through the antecubital vein catheter over 20 s, and a PET scan was performed to measure MBF. Participants underwent a 6-h b-OH-B infusion (prime dose was 1.5 mg/kg/min for 20 min followed by constant rate of 0.75 mg/kg/min) or 6-h NaHCO3 infusion. At 280 min after the start of b-OH-B or NaHCO3 in- fusions, 15O-H2O was injected for repeated measurement of MBF. At 300 min, 18F-FDG ) was injected, followed by a dynamic PET scan for the measurement of MGU.
Time Frame: MGU after B-OH-B or NaHCO3 infusion for 6 hours at minute 360 minutes
Population: Only participants in group II (12 subjects) underwent the cardiac PET with B-OH-B and NaHCO3 infusion , not in groups I and III
Measure: Mean (Standard Deviation); unit: µmol/ (min x 100 g)
Groups:
- Group I Beta-Hydroxy-Butyrate: There were no participants included in this outcome from Group I
- Group III Beta-Hydroxy-Butyrate: There were no participants in this group that were included in this outcome
Arm/Group | Group II Beta-Hydroxy-Butyrate | Group I Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Number analyzed (Participants) | 12 | 0 | 0
µmol/ (min x 100 g)
  Beta -H-B infusion | 9.6 (1.01) |  |
  NaHCO3 infusion | 8.56 (0.74) |  |

5. Secondary Outcome: Myocardial Energetics- Myocardic Blood Flow (MBF)
Description: as for outcome 4
Time Frame: MBF after B-OH-B or NaHCO3 infusion for 6 hours at 360 minutes (the results showed the difference betweenB-OH-B and NaHCO3 infusion for 6 hours)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
Number analyzed (Participants) | 0 | 12 | 0
ml/min |  | 0.05 (0.10) |

ADVERSE EVENTS:
Time Frame: From enrollment until end of study procedures at 360 minutes
Arm/Group | Group I Beta-Hydroxy-Butyrate | Group II Beta-Hydroxy-Butyrate | Group III Beta-Hydroxy-Butyrate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03560323/Prot_SAP_000.pdf